CLINICAL TRIAL: NCT02281006
Title: Randomized Controlled Trial to Test the Efficacy of Trans-tympanic Injections of a Sodium Thiosulfate Gel to Prevent Cisplatin-induced Ototoxicity in Patients With Head and Neck Cancer
Brief Title: Efficacy of Trans-tympanic Injections of a Sodium Thiosulfate Gel to Prevent Cisplatin-induced Ototoxicity
Acronym: STS001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, François Meyer, Researcher, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A13-09-985
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: DDP; Head and Neck Cancer; Adverse Effect
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated ear (Experimental): Trans-tympanic injection of a sodium thiosulfate gel
  Interventions: Drug: Trans-tympanic injection of a sodium thiosulfate gel
- Control ear (No Intervention): No intervention

INTERVENTIONS:
Drug: Trans-tympanic injection of a sodium thiosulfate gel — A sodium thiosulfate hyaluronate gel will be prepared by mixing 0.55 ml of a 25% solution of sodium thiosulfate pentahydrate (Seacalphyx, DIN 02386666, Seaford Pharmaceuticals Inc.) and 0.55 ml of a hyaluronate gel (Healon 10 mg, Abbott Medical Optics Inc.). On the day before each Cisplatin treatment an otologist will deposit 0.1 ml of the gel exactly on the round window of the middle ear.
  Other Names: Seacalphyx
  Arms: Treated ear

SUMMARY:
This study evaluates whether a gel containing sodium thiosulfate deposited via a trans-tympanic injection on the round window of the middle ear could reduce the ototoxicity caused by the drug Cisplatin among patients with head and neck cancer treated by chemoradiation. One ear selected randomly will be treated while the other will serve as control.

DETAILED DESCRIPTION:
Background

Cisplatin (cis-DiammineDichloridoPlatinum, DDP) is an antineoplastic agent used in the treatment of solid malignant tumors in adults and is also a key part of treatment for many children and adolescents with cancer. However, treatment with Cisplatin carries the risk of serious dose-limiting adverse effects. Ototoxicity is of major concern since the associated hearing loss greatly impairs patients' quality of life and no preventive treatment is presently available. Cisplatin ototoxicity is an important problem for patients treated for head and neck squamous cell carcinoma (HNSCC) who receive repeatedly high doses.

Cisplatin causes an accumulation of reactive oxygen species (ROS) in the cochlea, triggering damage to the outer hair cells of the organ of Corti. Sulfur-containing antioxidants can neutralize ROS following Cisplatin intoxication, and thus represent a potential preventive measure. A few sulfur-containing molecules have been studied. Experimental and human studies have shown that sodium thiosulfate (STS) can protect against Cisplatin-induced ototoxicity. However, when administered through the blood stream, STS interfere with Cisplatin treatment efficacy. To counter the ototoxic effects of Cisplatin treatment without impairing its efficacy, a local pharmacology approach directly aiming at the cochlea, would represent a powerful clinical strategy.

The proposed study is the first to test the efficacy of STS administered locally in the middle ear to prevent Cisplatin-induced ototoxicity in humans.

Objective

The objective of this study is to test the efficacy of trans-tympanic injections of a sodium thiosulfate-hyaluronate gel prior to cisplatin treatments to prevent cisplatin-induced ototoxicity in patients with locally advanced head and neck cancer.

The principal objective is to test the efficacy of the trans-tympanic injections of the gel at pure tone high frequencies. Exploratory analyses for secondary objectives will assess 1) cochlear damage, specifically hair cell function and 2) hearing loss at frequencies used for speech perception. Other outcomes considered are the severity of ototoxicity and the adverse effects of the trans-tympanic injections.

Methods

The proposed study is a randomized controlled trial. For each participant, one randomly selected ear will receive the treatment while the other ear will not. For ethical reasons, the control ear will not receive a placebo injection.

Participants to the trial will be recruited at the radiation therapy department of the CHU de Québec. Eligible participants are patients newly diagnosed with a locally advanced squamous cell carcinoma of the head and neck scheduled to be treated with concomitant chemoradiation. This treatment includes Cisplatin 100 mg/m2 on days 1, 22, and 43 after the first radiation fraction.

At the end of the first day of radiation therapy, the pharmacy department of the CHU de Québec will prepare the sodium thiosulfate hyaluronate gel by mixing 0.55 ml of a 25% solution of sodium thiosulfate pentahydrate (Seacalphyx, Drug identification number (DIN) 02386666, Seaford Pharmaceuticals Inc.) and 0.55 ml of a hyaluronate gel (Healon 10 mg, Abbott Medical Optics Inc.). After a local anesthesia of the tympanic membrane, the otologist will deposit 0.1 ml of the gel exactly on the round window of the middle ear. From there the STS should diffuse towards the cochlea. The same procedure will be repeated on the eve of the subsequent Cisplatin treatments on days 22 and 43.

To assess the effect of the trial intervention, a complete audiologic evaluation will be conducted before and one month after the end of chemoradiation therapy. The CHU de Québec audiologists will perform audiograms at frequencies ranging from 0.5 to 14 kHz. Sound intensity will be measured as dBHL(decibel hearing level). Speech reception thresholds will also be assessed. In addition, distortion product otoacoustic emissions (DPOAEs) recording will also be performed. Otoacoustic emissions measurements could detect hair cell damage due to Cisplatin early. The final audiologic evaluation will be conducted by an audiologist blinded to the ear assignment who would not have access to the trial and hospital records.

Adverse effects of the transtympanic injection will be documented according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE). In addition, to identify unexpected adverse effects of the trial intervention on hearing, a shorter unblinded audiogram will be conducted before proceeding to the second and third transtympanic injections. Data from these audiograms will not be used in the main analysis.The follow-up for audiologic safety monitoring will be continued for one year after the end of the trial.

The principal outcome is the hearing loss defined by the difference between the average permanent threshold shift (PTS) in dB (decibel) at four pure tone high frequencies (9, 10, 12.5 and 14 kHz) using the data from the audiograms done before and after Cisplatin therapy, for each patient and for each ear. The average PTS in dB at these pure tone high frequencies will be compared between the treated and the control ears using a t-test for paired data. A planned interim analysis will be conducted when half of the anticipated participants would have completed the follow-up. In the interim analysis, the test for superiority will be done with two-sided alpha=0.01 and the results shown only to the Data and Safety Monitoring Committee (DSMC). If the DSMC recommendation is to continue the trial as planned, the final analysis will be done with two-sided alpha=0.045 in order to keep the trial overall statistical significance level to 0.05.

Exploratory analyses for secondary outcomes will assess 1) cochlear damage, specifically hair cell function obtained from the results of DPOAEs, ands 2) the difference between the PTS in dB at pure tone averages (0.5 to 8 kHz), which represent frequencies for speech perception. Other outcomes considered are ototoxicity severity according to CTCAE, and adverse effects of the transtympanic injections.

The investigators have established an independent DSMC to overview the conduct of the trial comprising experts in biostatistics, audiology, and haemato-oncology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed locally advanced (stage III or IV) squamous cell carcinoma of the mouth, oropharynx, hypopharynx, or larynx scheduled to be treated with concomitant chemoradiation including Cisplatin100 mg/m2 3 times
* Normal otoscopic findings and symmetrical hearing

Exclusion Criteria:

* Karnofsky below 70

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Hearing loss at high frequencies | One month after Cisplatin treatment
  Hearing loss defined by the difference between the average permanent threshold shift (PTS) in dB (decibel) at four pure tone high frequencies (9, 10, 12.5 and 14 kHz) using the data from the audiograms done before and one month after Cisplatin therapy, for each patient and for each ear.

SECONDARY OUTCOMES:
Cochlear damage | One month after Cisplatin treatment
  Cochlear damage defined by the difference between the distortion product otoacoustic emissions (DPOAEs) recording before and one month after Cisplatin therapy, for each patient and for each ear.
Hearing loss at lower frequencies | One month and one year after Cisplatin treatment
  Hearing loss defined by the difference between the average permanent threshold shift (PTS) in dB (decibel) at four pure tone frequencies (0.5 to 8 kHz) using the data from the audiograms done before and one month and one year after Cisplatin therapy, for each patient and for each ear.
Adverse effects of trans-tympanic injections | One month after Cisplatin treatment
  Ototoxicity severity according to CTCAE after each trans-tympanic injection

CONTACTS AND LOCATIONS:
Overall Officials: Francois Meyer, MD, DSc, Principal Investigator — CHU de Quebec (Université Laval)
Locations (1):
- CHU de Quebec, Québec, Quebec, Canada